CLINICAL TRIAL: NCT01638403
Title: Randomized, Double-blind, Placebo and Comparator-controlled, Parallel-group, Multi-center Trial Assessing the Effects of BF2.649 in the Treatment of Excessive Daytime Sleepiness in Narcolepsy
Brief Title: Effects of BF2.649 in the Treatment of Excessive Daytime Sleepiness in Narcolepsy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bioprojet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P09-15/ BF2.649 Harmony 1bis
Record Dates: First submitted 2012-07-09; First posted 2012-07-11 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Treatment of Excessive Daytime Sleepiness in Narcolepsy
Keywords: narcolepsy; excessive daytime sleepiness; cataplexy
MeSH Terms: conditions — Narcolepsy; Disorders of Excessive Somnolence; Cataplexy | interventions — pitolisant; FANG vaccine; Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BF2.649 (Experimental): BF2.649 (pitolisant) is a novel, highly potent, selective, orally active histamine H3 receptor antagonist/inverse agonist (Ki of 0.3 nM) at the human receptor.
  Interventions: Drug: BF2.649
- Vigil (Active Comparator): Therapeutic indications Narcolepsy with and without cataplexy. Moderate to severe obstructive sleep apnoea syndrome with excessive daytime sleepiness despite adequate CPAP therapy.
  Moderate to severe chronic shift work sleep disorder with excessive sleepiness in patients who work rotating night shifts, if other sleep hygiene measures did not lead to a satisfactory improvement.
  Interventions: Drug: Vigil
- Placebo (Placebo Comparator)
  Interventions: Drug: palcebo

INTERVENTIONS:
Drug: BF2.649 — BF2.649 is provided in capsules. One-quarter or one-half of BF2.649 tablet at 20 mg (corresponding to 5-, and 10 mg, respectively).
  Patients should take 2 capsules per day with a glass of water. They will be instructed to take 1 capsule in the morning (after waking up, before breakfast around 8.00 a.m.) and 1 capsule at noon.
  Other Names: Pitolisant
  Arms: BF2.649
Drug: Vigil — Modafinil is provided in capsules. The capsules are identical in appearance to ensure that neither the patient nor the investigator nor members of the clinical staff knows the identity of the study medication.
  Modafinil tablet at 100 mg are enclosed in gelatine capsules. Patients should take 2 capsules per day with a glass of water. They will be instructed to take 1 capsule in the morning (after waking up, before breakfast around 8.00 a.m.) and 1 capsule at noon.
  Other Names: Modafinil
  Arms: Vigil
Drug: palcebo — placebo is provided in capsules. The capsules are identical in appearance to ensure that neither the patient nor the investigator nor members of the clinical staff knows the identity of the study medication.
  placebo consist of identical capsules containing lactose only. Patients should take 2 capsules per day with a glass of water. They will be instructed to take 1 capsule in the morning (after waking up, before breakfast around 8.00 a.m.) and 1 capsule at noon.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
3. RATIONALE FOR BF2.649 IN NARCOLEPSY Narcolepsy is a disabling syndrome affecting the generation and organizations of sleep and wakefulness, first described by Westphal and Gelineau in 19th century. Excessive Daytime Sleepiness (EDS) and cataplexy are two main symptoms of narcolepsy. Other symptoms referred to as auxiliary symptoms are hypnagogic and hypnopompic hallucinations, sleep paralysis, dyssomnia and automatic behaviour. The prevalence of narcolepsy is estimated around 25 per 100 000 in Causasian population. It is often extremely incapacitating, interfering with every aspect of life, in work and social settings.

Several breakthroughs in the understanding of physiopathology of narcolepsy have recently shown that most narcoleptic patients display a strongly decreased CSF level of orexins, a group of hypothalamic peptides with wake-promoting activity. It was also found that sporadic narcolepsy in dogs, mice and humans may also be related to a deficiency in the production of orexin ligands. Narcolepsy may be a neurodegenerative or autoimmune disorder resulting in a loss of hypothalamic neurons containing the orexin [Baumann CR & Bassetti CL Lancet Neurol. 2005 ; Dauvilliers Y et al, Clin Neurophysiol. 2003 ].

In accordance with guidelines published by the European task force [Billiard M et al, Eur J Neurol. 2006] , management of narcolepsy with or without cataplexy relies on several classes of drugs, namely stimulants for EDS, antidepressants for cataplexy and hypnosedative drugs for disturbed nocturnal sleep. The first line pharmacological treatment of EDS and irresistible episodes of sleep rely on Modafinil, 100-400 mg/day, given in two doses, one in the morning and one early in the afternoon, the need for amphetamines and amphetamine-like stimulants (e.g. methylphenidate) has been decreased. Sodium oxybate and antidepressants are main drug therapies of cataplexy.

BF2.649, an H3R inverse agonist promotes significantly vigilance in mice knock out for the orexin gene, a reliable model of narcolepsy, whereas the animals remain calm, a difference with treatment by amphetamine-like drugs which induce psychomotor excitation. In addition, BF2.649 shows a significant inhibitory effect on the occurrence of narcolepsy episodes during the dark period. These narcolepsy episodes are to be compared to cataplexy episodes in human [Chemelli et al., Cell 1999] 11. In agreement, Modafinil, in humans, does not show any effects on cataplexy, even if it improves wakefulness by an ill-defined mechanism. Thus anticataplectic drugs, such as antidepressants, are given in addition to Modafinil to narcoleptic patients.

Taken together, the preclinical and clinical results provide a compelling rationale for this study to verify and confirm, under randomized double-blind and placebo-controlled conditions, the safety and efficacy of escalating dose of BF2.649 in the treatment of EDS and cataplexy in narcolepsy.

It is on the basis of preclinical studies, and on the observation of the first included patients, that the doses to be administered were determined.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females of any ethnic origin, 18 years old and over.
2. Both new and previously diagnosed patients with narcolepsy with or without cataplexy could be included. All patients should meet the International Classification of Sleep Disorders (ICSD-2) criteria.
3. Patients should be free of drugs or discontinue any psychostimulant medications for at least 14 days at the start of baseline period. Patients with severe cataplexy are permitted to remain on their anticataplectic medication at stable dose except tricyclic antidepressants. The authorized anticataplectic treatment should have been administrated for at least 1 month prior to the trial and these doses should not be changed throughout the trial (from V1 to V8).
4. Epworth Sleepiness Scale (ESS) score should be ≥ 14 during the baseline period.
5. Patients have expressed a willingness to participate in and complete the study, and signed and dated informed consent prior to beginning protocol required procedures.
6. Females must be surgically sterile or 2 years postmenopausal. Females of child-bearing potential must use a medically accepted effective method of birth control (i.e. oral contraceptives of normal average dosage ≥ 0.05 mg ethinyl-oestradiol, intra-uterine device, with a barrier method such as spermicides…), agree to continue this method for the duration of the study and be negative to serum pregnancy test performed at the screening visit. Females should not be breast-feeding patient.
7. In the opinion of the investigator, the patient must have adequate support to comply with the entire study requirements as described in the protocol (e.g., transportation to and from trial site, self rating scales and diaries completion, drug compliance, scheduled visits, tests).
8. If indicated by investigator, the patient must be willing to not operate a car or heavy machinery for the duration of the trial or as long as the investigator deems clinically indicated. In addition, the patient should be willing to maintain during the study their usual behaviour which could affect their diurnal sleepiness (e.g. circadian rhythm, caffeine consumption, nocturnal sleep duration).
9. Patient should be assured by appropriate healthy insurance system (only applicable where mandatory e.g. in France).

Exclusion Criteria:

1. The use of BF2.649 or any previous investigational drugs within 30-day period prior to initial screening visit (V1) for this trial.
2. In narcoleptic patients without cataplexy, they should not have any other conditions that can be considered the primary causes of EDS: such as sleep related breathing disorders as defined by a sleep Apnea Index ≥ 10 per hour or and an Apnea/Hypopnea Index ≥ 15 per hour, periodic limbs movement (PLM) disorders as defined by a PLM arousal index (PLMAI) ≥ 10 per hour, shift work, chronic sleep deprivation, circadian sleep wake rhythm disorder or any other medical or neurological causes that could account for narcolepsy symptoms associated with EDS.
3. Patients who are unable or unwilling to temporarily discontinue any no-authorized drugs or substances (see Section Non-authorized treatments).
4. Current or recent (within one year) history of a substance abuse or dependence disorder including alcohol abuse as defined in Diagnostic and Statistical Manual of Mental Disorders (DSM-IV).
5. Any significant serious abnormality of the cardiovascular system e.g. recent myocardial infarction, angina, hypertension or dysrhythmia (within the prior 6 months), Electrocardiogram Bazett's corrected QT interval (QT x square root[HR/60]) higher than 450 ms, history of left ventricular hypertrophy or mitral valve prolapse.
6. Patients with severe depression (BDI13 ≥ 16) or with a suicidal risk (item G BDI13 > 0)
7. Patients with Severe hepatic Impairment (e.g. prothrombin ratio, < 50% or factor V < 50% if the patient receiving anti-vitamin K) or with Severe Renal Impairment (e.g. serum creatine greater than 2.0 mg/dL), or with any other significant abnormality in the physical examination or clinical laboratory results.
8. Psychiatric and neurological disorders, such as moderate or severe psychosis or dementia, bipolar illness, severe anxiety, clinical depression, history of seizure disorder or other problem that in the investigator's opinion would preclude the patient's participation and completion of this trial or comprise reliable representation of subjective symptoms.
9. Prior severe adverse reactions to CNS stimulants.
10. Known hypersensitivity to the tested treatment including active substance and excipients.
11. The inability to continue daily activities safely, without the use of treatment against EDS.
12. Other active clinically significant illness, including unstable cardiovascular, endocrine, neoplastic, gastrointestinal, hematologic, hepatic, immunologic, metabolic, neurological (other than narcolepsy/cataplexy), pulmonary, and/or renal disease which could interfere with the study conduct or counter-indicate the study treatments or place the patient at risk during the trial or compromise the study objectives.
13. Any patients presenting congenital galactosemia, glucose-galactose malabsorption or lactase deficiency due to the presence of lactose in investigational treatments
14. Patients participating in another study or being in a follow-up period for another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2010-11; Primary Completion 2012-04 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Epworth Sleepiness Scale scores (ESS) | 10 weeks
  The primary efficacy endpoint is Epworth Sleepiness Scale scores (ESS) change between the BF2.649-treatment group, the placebo-group, and the Modafinil-treatment group during an 8-week treatment period.
  The ESS is a self-administered questionnaire to the patients to evaluate their chances of dozing in height different situations often encountered in the daily life.
  The average of ESS performed at V6 and V7 will be compared to the average of ESS performed at V2 and V3.

SECONDARY OUTCOMES:
patient sleep diary | 10 weeks
  Following secondary outcome measures will be reported in the patient sleep diary:
  1. Number and duration of diurnal involuntary sleep attacks and episodes of severe sleepiness
  2. Number of cataplexy total and partial.
  3. Number of hallucinations.
  4. Number of sleep paralysis.
  5. Number and duration of nocturnal awakening and total duration of nocturnal sleep time.
Maintenance of Wakefulness Test (MWT) | 10 weeks
  The Maintenance of Wakefulness Test (MWT) is used in this study to assess an individual's ability to maintain awake while resisting the pressure to fall asleep. Patients will be administrated four 40-minute MWT sessions at 2 hours interval at inclusion visit (V3) and at endpoint visit (V7 or the last on-study visit), according to validated standard [Doghramji K et al, Electroencephalogr Clin Neurophysiol. 1997] . The changes in MWT will be compared between the treatment groups. The MWT will be renewed at V7 only for patients who had a MWT <11 at V3.
Test of Sustained Attention to Response Task (SART) | 10 weeks
  The Test of Sustained Attention to Response Task (SART) has been used for the quantification of vigilance and attention in narcolepsy patients [Fronczek R et al, Sleep 2006] . The SART will be performed at inclusion visit (V3) and at endpoint (V7 or the last on-study visit for prematurely withdrawn patients). The changes in SART will be compared between the treatment groups.
Clinical Global Impressions of Change | 10 weeks
  The severities of EDS and of cataplexy will be measured at baseline by the investigator using the Clinical Global Impression of Severity (CGI-S) in order to describe the population. At each follow-up visit, the patients' change in EDS and in cataplexy compared to baseline will be rated by the same investigator using Clinical Global Impression of Change (CGI-C) to document the perceived change in patients' illness.
European Quality of life questionnaire (EQ-5D) | 10 weeks
  EQ-5D is a reliable and validated measure of quality of life. Narcolepsy has a clear negative effect on this outcome measure [Dodel R. et al, Sleep Med. 2007] . EQ-5D will be completed at baseline visit (V2), inclusion visit (V3), stable-dose visit (V5), endpoint visit (V7) and withdrawal visit (V8). The changes between treatment groups will be analysed as an evaluation of the illness evolution.
Patient's Global Opinion on the effect of treatment | 10 weeks
  At each visit under treatment (V4, V5, V6, V7 and V8 or last on-study visit), patients evaluate the Global effect of their treatment by comparing the period prior to that visit with the patient's prestudy condition.

CONTACTS AND LOCATIONS:
Overall Officials: DAUVILLIERS Yves, Study Chair — Hôpital Gui de Chauliac - 80, avenue A. Fliche , 34295 Montpellier cedex 5 - FRANCE
Locations (1):
- Evelyne DESCHAMPS DE PAILLETTE, Paris, France

REFERENCES:
- [Background] Fronczek R, Middelkoop HA, van Dijk JG, Lammers GJ. Focusing on vigilance instead of sleepiness in the assessment of narcolepsy: high sensitivity of the Sustained Attention to Response Task (SART). Sleep. 2006 Feb;29(2):187-91. PMID 16494086
- See also: Related Info — http://www.bioprojet.com